CLINICAL TRIAL: NCT04522102
Title: An Investigator Initiated and Conducted, Prospective, Multicentre, Randomised Outcome-blinded Pilot Study of Antiplatelet Therapy in Patients with a History of Stroke Due to Intracerebral Haemorrhage
Brief Title: Antiplatelet Secondary Prevention International Randomised Trial After INtracerebral HaemorrhaGe (ASPIRING)-Pilot Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: University of Edinburgh (Other); Huashan Hospital (Other); The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASPIRING
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: stroke; intracerebral hemorrhage; antiplatelet therapy; aspirin; clopidogrel; cilostazol
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Start antiplatelet monotherapy (one antiplatelet drug available in local standard clinical practice, chosen by patient's physician pre-randomisation).
  Interventions: Drug: Start antiplatelet monotherapy
- Comparator (No Intervention): Avoid antiplatelet therapy.

INTERVENTIONS:
Drug: Start antiplatelet monotherapy — Start one antiplatelet drug, be available in local standard clinical practice, chosen by patient's physician pre-randomisation
  Arms: Intervention

SUMMARY:
ASPIRING is an investigator-led, multicentre, prospective, randomised, open-label, blind outcome (PROBE), parallel group, clinical trial. The pilot phase will explore the feasibility of conducting a trial of starting antiplatelet monotherapy versus avoiding antiplatelet therapy for reducing all serious vascular events for adults surviving symptomatic stroke due to spontaneous intracerebral haemorrhage (ICH). The pilot phase will involve ~120 patients at ~30 hospitals in China, Australia and New Zealand.

DETAILED DESCRIPTION:
The participant eligibility criteria specifically identify adults with history of symptomatic spontaneous ICH. Randomisation occurs if a participant and their doctor are uncertain about whether to start or avoid antiplatelet monotherapy at least 24 hours after ICH symptom onset. The intervention is a pragmatic policy of starting antiplatelet monotherapy (one antiplatelet drug available in local standard clinical practice, chosen by patient's physician pre-randomisation). The control group adopts a policy of avoiding antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18 years.
2. Symptomatic stroke due to spontaneous (non-traumatic) ICH.
3. Patient is at least 24 hours after ICH symptom onset.
4. Patient and their doctor are both uncertain about whether to start or avoid antiplatelet monotherapy.
5. Consent to randomisation from the patient (or personal / legal / professional representative if the patient does not have mental capacity).

Exclusion Criteria:

1. ICH due to head injury, in the opinion of the investigator.
2. ICH due to haemorrhagic transformation of an ischaemic stroke, in the opinion of the investigator.
3. Patient is already taking antiplatelet therapy, or full dose anticoagulant therapy, after ICH.
4. Patient is pregnant, breastfeeding, or of childbearing age and not taking contraception.
5. Patient and carer unable to understand spoken or written local language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
regulatory approvals | 6 months
  Receipt of regulatory approvals in China，Australia and New Zealand separately, including Ethics, Human Genetics Resources Administration of China (HGRAC).

SECONDARY OUTCOMES:
trial database | 6 months
  Trial database structure and data flows that comply with data privacy and information governance regulations in China, Australia and New Zealand.
Site recruitment | 12-18 month
  Participation of 20 sites in China and 10 sites in Australia and New Zealand
Calculate frequency of clinical data | 3 years
  Frequency of ICH survivors who are screened, eligible, approached, consented, and randomised by month and site from activation.
Barriers to randomisation of eligible patients. | 3 years
  Barriers to randomisation of eligible patients.
Frequency of protocol deviations and violations. | 3 years
  Frequency of protocol deviations and violations.
Adherence to the allocated intervention by investigators and participants | 3 years
  Adherence to the allocated intervention by investigators and participants
Frequency of withdrawal and loss to follow-up | 3 years
  Frequency of withdrawal and loss to follow-up
Completeness of follow-up assessments | 3 years
  Completeness of follow-up assessments
Characteristics of randomised participants compared with eligible patients who were not recruited. | 3 years
  Characteristics of randomised participants compared with eligible patients who were not recruited.
Frequency of the composite of all serious vascular events | 6 months
  composite of all serious vascular events (non-fatal stroke, non-fatal myocardial infarction or death from a vascular cause)
Serious adverse event (SAE) | at least 6 months
  any serious adverse event (SAE)
Serious adverse reaction (SAR) | at least 6 months
  serious adverse reaction (SAR)
Suspected Unexpected Serious Adverse Reaction (SUSAR) | at least 6 months
  Suspected Unexpected Serious Adverse Reaction (SUSAR)

CONTACTS AND LOCATIONS:
Overall Officials: Rustam Al-Shahi Salman, Principal Investigator — University of Edinburgh; Craig S Anderson, Principal Investigator — The George Institute; Graeme Hankey, MD, Principal Investigator — The University of Western Australia
Locations (2):
- China (2):
  - The George Institute for Global Health, Beijing, Beijing Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170
- [Derived] Cheng X, Dong Q. Towards individualised secondary prevention after intracerebral haemorrhage. Lancet Neurol. 2021 Jun;20(6):411-413. doi: 10.1016/S1474-4422(21)00130-7. No abstract available. PMID 34022160